CLINICAL TRIAL: NCT02821169
Title: Impact of Infiltration in the Region of the Palatine Ganglion Spheno by Ropivacaine on Postoperative Pain in the Setting of Endoscopic Sinonasal Surgery.
Brief Title: Infiltration in the Region of the Palatine Ganglion Spheno by Ropivacaine on Postoperative Pain
Acronym: ROPI_POSTOP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013_07; 2013-004410-17 (EudraCT Number)
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2019-09

CONDITIONS: Pain
Keywords: sinus surgery; sphenopalatin ganglion; ropivacaine; local anesthesia
MeSH Terms: conditions — Pain | interventions — Ropivacaine; Saline Solution; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- saline solution 0.9% (Placebo Comparator): injection of saline solution in the sphenopalatine area in both nasal fossa
  Interventions: Drug: saline solution 0.9%
- ropivacaine (2mg/ml) (Active Comparator): injection of ropivacaine in the sphenopalatine area in both nasal fossa
  Interventions: Drug: ropivacaine

INTERVENTIONS:
Drug: ropivacaine — injection of 4mL of ropivacaine in the sphenopalatine area through an endoscopic approach
  Other Names: NAROPEINE
  Arms: ropivacaine (2mg/ml)
Drug: saline solution 0.9% — injection of 4 mL of saline solution in the sphenopalatine area through an endoscopic approach
  Other Names: NaCL 0.9% injectable
  Arms: saline solution 0.9%

SUMMARY:
Endoscopic sinus surgery (ESS) is a prevalent surgical procedure. It is required in many chronic rhinosinusitis for whom the medical treatment failed. In order to improve the postoperative management of patients treated with ESS, we aim to assess the analgesic action of local injection of ropivacaine in the nasal fossa.

DETAILED DESCRIPTION:
A prospective randomized double blind placebo controlled study was designed. Local injection of ropivacaine or placebo was conducted at the end of the surgical procedure in both nasal fossa through endoscopic view in the sphenopalatine region.

Pain was measured in the postoperative course with visual analogic scale in the recovery room and the rhinologic department.

ELIGIBILITY:
Inclusion Criteria:

* patients requiring endoscopic sinus surgery
* ASA score 1 or 2
* patients with health care insurance
* approved consent

Exclusion Criteria:

* any sinonasal malignant tumor
* renal failure, hepatic disorder, respiratory deficiency, cardiovascular diseases
* neurologic disorders
* alcohol or drugs addiction
* preoperative facial pain from an extranasal origin
* coagulation disorders
* antidepressive treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | at the 2 postoperative hours
  Measure the intensity pain, in the group treated with Ropivacaine.

SECONDARY OUTCOMES:
Analgesics consumption orally | during the 7 days post-surgery
  patient-controlled administration
Administration of analgesics by parenteral route | at the 2 postoperative hours
  patient-controlled administration
Visual analog scale for the intensity postoperative pain | at the 4 and at the 6 postoperative hours
  patient-controlled administration
Visual analog scale for the during postoperative pain | At Morning and evening between the 1 and 7 days post surgery
  self-assessment by the patient at home on the information collection book

CONTACTS AND LOCATIONS:
Overall Officials: Goeffrey Mortuaire, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHRU, Hôpital Claude Huriez, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Morisse M, Rysman B, Szymanski C, Fackeure R, Mouawad F, Mortuaire G. A randomized placebo-controlled trial assessing sphenopalatine ganglion block in endoscopic sinus surgery. Int Forum Allergy Rhinol. 2021 Sep;11(9):1384-1386. doi: 10.1002/alr.22804. Epub 2021 May 19. No abstract available. PMID 34013619